CLINICAL TRIAL: NCT01886040
Title: Factors Affecting the Prognosis of Patients With Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 102058-E
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-02

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- cases with endometrial cancer

SUMMARY:
Endometrial cancer is the second common gynecologic malignancy in Taiwan. The prevalence has been overcome the epithelial ovarian cancer because of the change of life style to western style recently. Most patients with endometrial cancer are stage I & II, the most histology is still "endometrioid adenocarcinoma" (type I endometrial cancer). In statistics, advanced stage (FIGO stage III and IV) is approximately 16% of all cases.

Most patients has good outcome of endometrial cancer because their surgical stage is belonged to "early stage". However, the recurrence, distant metastases and mortality are high if the diseases is confirmed to be advanced stage. The adjuvant therapies after staging/debulking operation are systemic chemotherapy and whole pelvic radiation therapy/ brachytherapy. Whether the adjuvant therapy can cure the disease of not is still controversial.

Because of the rarity of the advanced endometrial cancer, varies adjuvant therapeutic modalities, eg. chemotherapy only, pelvic radiation therapy only, combination of chemotherapy and radiation therapy or sequential "sandwich" therapy were ever used for such group patients in each medical center. But the case number is insufficient and limited to show the survival or progression free benefit during the statistics. Besides, the surgical procedures and adjuvant therapy for early endometrial cancer is still remained to be determined. The investigators are also interested to analyze the factors affecting their survival.

The investigators will perform a retrospective study to review the data of patients with endometrial cancer in Department of Obstetrics & Gynecology in Far Eastern Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Time interval: from 1991 to date.
2. Comprehensive surgical staging or debulking procedure.
3. All female patients with endometrial cancer who underwent surgery for endometrial cancer at Far Eastern Memorial Hospital.

Exclusion Criteria:

1. Not comprehensive staging/debulking procedure.
2. Patients who died of postoperative complications within 30 days after surgery were excluded from the survival analysis.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the cases with endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Factors affecting overall survival and disease-free survival of endometrial cancer | 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan